CLINICAL TRIAL: NCT01958671
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, 26-week Multicenter Study With a 26-Week Extension to Evaluate the Efficacy and Safety of Ertugliflozin Monotherapy in the Treatment of Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control Despite Diet and Exercise
Brief Title: A Study of the Efficacy and Safety of Ertugliflozin Monotherapy in the Treatment of Participants With Type 2 Diabetes Mellitus and Inadequate Glycemic Control Despite Diet and Exercise (MK-8835-003, VERTIS MONO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-003; 2013-002519-90 (EudraCT Number); B1521022 (Other: Pfizer Protocol Number)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ertugliflozin 5 mg/Ertugliflozin 5 mg (Experimental): Phase A: Ertugliflozin 5 mg administered once daily for 26 weeks. Participants requiring rescue therapy will receive open-label metformin. Phase B: Ertugliflozin 5 mg administered once daily for 26 weeks. Participants not rescued with metformin in Phase A, will receive placebo to metformin. Participants rescued with metformin in Phase A will continue to receive metformin. Participants requiring rescue therapy during Phase B will receive open-label glimepiride.
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo to Ertugliflozin; Drug: Metformin; Drug: Placebo to Metformin; Drug: Glimepiride
- Ertugliflozin 15 mg/Ertugliflozin 15 mg (Experimental): Phase A: Ertugliflozin 15 mg administered once daily for 26 weeks. Participants requiring rescue therapy will receive open-label metformin. Phase B: Ertugliflozin 15 mg administered once daily for 26 weeks. Participants not rescued with metformin in Phase A, will receive placebo to metformin. Participants rescued with metformin in Phase A will continue to receive metformin. Participants requiring rescue therapy during Phase B will receive open-label glimepiride.
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Ertugliflozin 10 mg; Drug: Metformin; Drug: Placebo to Metformin; Drug: Glimepiride
- Placebo/Metformin (Other): Phase A: Placebo to ertugliflozin administered once daily for 26 weeks. Participants requiring rescue therapy will receive open-label metformin. Phase B: Participants not rescued with open-label metformin in Phase A will also receive blinded metformin up to twice daily for 26 weeks in addition to placebo. Participants rescued with metformin in Phase A will continue to receive open-label metformin. Participants requiring rescue therapy during Phase B will receive open-label glimepiride.
  Interventions: Drug: Placebo to Ertugliflozin; Drug: Metformin; Drug: Glimepiride

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — One tablet taken orally the same time in the morning from Day 1 through Week 52 (Phase A and Phase B).
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 15 mg/Ertugliflozin 15 mg; Ertugliflozin 5 mg/Ertugliflozin 5 mg
Drug: Ertugliflozin 10 mg — One tablet taken orally the same time in the morning from Day 1 through Week 52 (Phase A and Phase B).
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 15 mg/Ertugliflozin 15 mg
Drug: Placebo to Ertugliflozin — One placebo tablet matching the ertugliflozin 5 mg tablet and/or 1 placebo tablet matching the ertugliflozin 10 mg tablet per day taken orally the same time in the morning from Day 1 through Week 52 (Phase A and Phase B).
  Arms: Ertugliflozin 5 mg/Ertugliflozin 5 mg; Placebo/Metformin
Drug: Metformin — 500 mg (1 tablet) in the morning and 500 mg (1 tablet) in the evening for 2 weeks, 1000 mg (2 tablets 500 mg) in the morning and 500 mg (1 tablet) in the evening for 2 weeks and 1000 mg (2 tablets 500 mg) in the morning and 1000 mg (2 tablets 500 mg) in the evening, thereafter.
  Other Names: Glucophage XR, Carbophage SR, Riomet, Fortamet, Glumetza, Obimet, Gluformin, Dianben, Diabex, Diaformin, Siofor and Metfogamma.
Drug: Placebo to Metformin — 1 tablet in the morning and 1 tablet in the evening for 2 weeks, 2 tablets in the morning and 1 tablet in the evening for 2 weeks and 2 tablets in the morning and 2 tablets in the evening, thereafter.
  Arms: Ertugliflozin 15 mg/Ertugliflozin 15 mg; Ertugliflozin 5 mg/Ertugliflozin 5 mg
Drug: Glimepiride — Dosing and titration of glimepiride as rescue therapy was determined by the investigator.

SUMMARY:
This trial will evaluate the efficacy and safety of ertugliflozin monotherapy in the treatment of participants with type 2 diabetes mellitus (T2DM) and inadequate glycemic control on diet and exercise. This trial consists of a run-in period of 3 to 11 weeks, a 26-week placebo-controlled treatment period (Phase A), and a 26-week active treatment period (Phase B). The primary hypotheses of the trial are that at Week 26, the mean reduction from baseline in hemoglobin A1c (A1C) for 15 mg ertugliflozin is greater than that for placebo and the mean reduction from baseline in A1C for 5 mg ertugliflozin is greater than that for placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM in accordance to American Diabetes Association guidelines
* Participants with no prior allowable oral anti-hyperglycemic agents (AHA) for at least 8 weeks prior to study participation or participants on a single allowable oral AHA at the start of study participation
* Participants on a single allowable AHA must be willing to discontinue this medication at the Screening Visit (S2) and remain off this medication for the duration of the trial. Allowable oral AHAs for discontinuation are metformin, sulfonylureas, dipeptidyl peptidase-4 (DPP-4) inhibitors, glinides or alpha-glucosidase inhibitors.

Exclusion Criteria:

* History of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional class III-IV heart failure within 3 months of study participation
* A clinically significant electrocardiogram abnormality
* A history of malignancy ≤5 years prior to study participation, except for adequately treated basal or squamous cell skin cancer or in situ cervical cancer
* A known hypersensitivity or intolerance to any sodium-glucose co-transporter 2 (SGLT2) inhibitor or metformin
* On a blood pressure or lipid altering medication that have not been on a stable dose for at least 4 weeks prior to study participation
* A surgical procedure within 4 weeks prior to study participation or planned major surgery during the trial
* Donation of blood or blood products within 6 weeks of study participation or plans to donate blood or blood products at any time during the trial
* Pregnant or breast-feeding, or is expecting to conceive during the trial, including 14 days following the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2013-10-09 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Terra SG, Focht K, Davies M, Frias J, Derosa G, Darekar A, Golm G, Johnson J, Saur D, Lauring B, Dagogo-Jack S. Phase III, efficacy and safety study of ertugliflozin monotherapy in people with type 2 diabetes mellitus inadequately controlled with diet and exercise alone. Diabetes Obes Metab. 2017 May;19(5):721-728. doi: 10.1111/dom.12888. Epub 2017 Feb 22. PMID 28116776
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Gallo S, Raji A, Calle RA, Pong A, Meyer C. The effects of ertugliflozin on beta-cell function: Pooled analysis from four phase 3 randomized controlled studies. Diabetes Obes Metab. 2020 Dec;22(12):2267-2275. doi: 10.1111/dom.14149. Epub 2020 Aug 27. PMID 32700393
- [Derived] Gallo S, Calle RA, Terra SG, Pong A, Tarasenko L, Raji A. Effects of Ertugliflozin on Liver Enzymes in Patients with Type 2 Diabetes: A Post-Hoc Pooled Analysis of Phase 3 Trials. Diabetes Ther. 2020 Aug;11(8):1849-1860. doi: 10.1007/s13300-020-00867-1. Epub 2020 Jul 9. PMID 32648108
- [Derived] Patel S, Hickman A, Frederich R, Johnson S, Huyck S, Mancuso JP, Gantz I, Terra SG. Safety of Ertugliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Seven Phase 3 Randomized Controlled Trials. Diabetes Ther. 2020 Jun;11(6):1347-1367. doi: 10.1007/s13300-020-00803-3. Epub 2020 May 5. PMID 32372382
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Wu L, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Efficacy and safety of ertugliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Aug;36(8):1277-1284. doi: 10.1080/03007995.2020.1760228. Epub 2020 May 13. PMID 32324082
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Patel S, Hickman A, Mancuso JP, Ellison MC, Gantz I, Terra SG. Efficacy and safety of ertugliflozin in Hispanic/Latino patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Jul;36(7):1097-1106. doi: 10.1080/03007995.2020.1760227. Epub 2020 May 13. PMID 32324065
- [Derived] Liu J, Patel S, Cater NB, Wu L, Huyck S, Terra SG, Hickman A, Darekar A, Pong A, Gantz I. Efficacy and safety of ertugliflozin in East/Southeast Asian patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2020 Apr;22(4):574-582. doi: 10.1111/dom.13931. Epub 2020 Jan 3. PMID 31797522
- [Derived] Liu J, Pong A, Gallo S, Darekar A, Terra SG. Effect of ertugliflozin on blood pressure in patients with type 2 diabetes mellitus: a post hoc pooled analysis of randomized controlled trials. Cardiovasc Diabetol. 2019 May 7;18(1):59. doi: 10.1186/s12933-019-0856-7. PMID 31064361
- [Derived] Aronson R, Frias J, Goldman A, Darekar A, Lauring B, Terra SG. Long-term efficacy and safety of ertugliflozin monotherapy in patients with inadequately controlled T2DM despite diet and exercise: VERTIS MONO extension study. Diabetes Obes Metab. 2018 Jun;20(6):1453-1460. doi: 10.1111/dom.13251. Epub 2018 Feb 23. PMID 29419917

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg/Ertugliflozin 5 mg | Ertugliflozin 15 mg/Ertugliflozin 15 mg | Placebo/Metformin
Started | 156 | 152 | 153
Completed | 137 | 128 | 121
Not Completed | 19 | 24 | 32
Not completed — Adverse Event | 1 | 1 | 5
Not completed — Death | 1 | 0 | 0
Not completed — Excluded medication | 0 | 0 | 1
Not completed — Hyperglycemia | 0 | 0 | 2
Not completed — Lost to Follow-up | 7 | 11 | 7
Not completed — Non-compliance with study drug | 1 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Study site terminated by sponsor | 1 | 0 | 1
Not completed — Participant moved | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg/Ertugliflozin 5 mg | Ertugliflozin 15 mg/Ertugliflozin 15 mg | Placebo/Metformin | Total
Number analyzed (Participants) | 156 | 152 | 153 | 461
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (11.4) | 56.2 (10.8) | 56.1 (10.9) | 56.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 62 | 71 | 200
  Male | 89 | 90 | 82 | 261
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] — Population: All randomized participants who received at least 1 dose of study treatment and had baseline A1C measurement.
  Percent
    number analyzed (Participants) | 155 | 151 | 153 | 459
    (all) | 8.16 (0.88) | 8.35 (1.12) | 8.11 (0.92) | 8.21 (0.98)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Population: All randomized participants who received at least 1 dose of study treatment and had baseline FPG measurement.
  mg/dL
    number analyzed (Participants) | 151 | 149 | 150 | 450
    (all) | 180.9 (48.5) | 179.1 (48.2) | 180.2 (45.8) | 180.1 (47.4)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.75m^2] | 88.5 (18.4) | 88.3 (18.0) | 86.2 (19.4) | 87.7 (18.6)
Body weight [Mean (Standard Deviation); unit: Kilograms] | 94.0 (25.4) | 90.6 (18.3) | 94.2 (25.2) | 92.9 (23.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In A1C at Week 26
Description: A1C is measured as percent. The change from baseline is the Week 26 A1C percent minus the Week 0 A1C percent. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study treatment and had a baseline A1C measurement or at least 1 post-randomization A1C measurement subsequent to at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Ertugliflozin 5 mg: Participants received ertugliflozin 5 mg once daily for 26 weeks.
- Ertugliflozin 15 mg: Participants received ertugliflozin 15 mg once daily for 26 weeks.
- Placebo: Participants received placebo to ertugliflozin once daily for 26 weeks.
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 151 | 153
Percent | -0.79 [-0.95 to -0.63] | -0.96 [-1.12 to -0.80] | 0.20 [0.02 to 0.37]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; Fixed effects for treatment, time, prior anti-hyperglycemic medication, baseline eGFR and the interaction of time by treatment; Difference in least squares means = -0.99, 95% CI 2-sided [-1.22 to -0.76]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -1.16, 95% CI 2-sided [-1.39 to -0.93]

2. Primary Outcome: Percentage of Participants Experiencing An Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. Data presented include data following the initiation of rescue therapy.
Time Frame: Up to 54 weeks (including 2 weeks following last dose)
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study treatment. Participants were classified according to randomized treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg/Ertugliflozin 5 mg | Ertugliflozin 15 mg/Ertugliflozin 15 mg | Placebo/Metformin
Number analyzed (Participants) | 156 | 152 | 153
Percentage of participants | 64.1 | 62.5 | 66.7
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg/Ertugliflozin 5 mg vs Placebo/Metformin; Test type: Superiority or Other; Difference in percentage = -2.6, 95% CI 2-sided [-13.1 to 8.1] — Based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg/Ertugliflozin 15 mg vs Placebo/Metformin; Test type: Superiority or Other; Difference in percentage = -4.2, 95% CI 2-sided [-14.8 to 6.6] — Based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg/Ertugliflozin 5 mg | Ertugliflozin 15 mg/Ertugliflozin 15 mg | Placebo/Metformin
Number analyzed (Participants) | 156 | 152 | 153
Percentage of participants | 4.5 | 3.9 | 6.5
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg/Ertugliflozin 5 mg vs Placebo/Metformin; Test type: Superiority or Other; Difference in percentage = -2.0, 95% CI 2-sided [-7.7 to 3.3] — Based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg/Ertugliflozin 15 mg vs Placebo/Metformin; Test type: Superiority or Other; Difference in percentage = -2.6, 95% CI 2-sided [-8.2 to 2.7] — Based on Miettinen & Nurminen method

4. Secondary Outcome: Change From Baseline in FPG at Week 26
Description: The change from baseline is the Week 26 FPG minus the Week 0 FPG. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study treatment and had a baseline FPG measurement or at least 1 post-randomization FPG measurement subsequent to at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 155 | 152 | 153
mg/dL | -33.96 [-39.85 to -28.06] | -43.44 [-49.39 to -37.49] | 0.57 [-6.02 to 7.16]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -34.53, 95% CI 2-sided [-42.76 to -26.29]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -44.01, 95% CI 2-sided [-52.28 to -35.74]

5. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: The change from baseline is the Week 26 body weight minus the Week 0 body weight. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study treatment and had a baseline body weight measurement or at least 1 post-randomization body weight measurement subsequent to at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 152 | 153
Kilograms | -3.18 [-3.72 to -2.63] | -3.58 [-4.13 to -3.02] | -1.42 [-2.02 to -0.81]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -1.76, 95% CI 2-sided [-2.57 to -0.95]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -2.16, 95% CI 2-sided [-2.98 to -1.34]

6. Secondary Outcome: Percentage of Participants With A1C <7% (<53 mmol/Mol) at Week 26
Description: A1C is measured as percent. Laboratory measurements were performed after an overnight fast ≥10 hours in duration. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 151 | 153
Percentage of participants | 28.2 | 35.8 | 13.1
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Fixed effects for treatment, prior antihyperglycemic medication, covariates for baseline A1C and baseline eGFR; Odds Ratio (OR) = 3.59, 95% CI 2-sided [1.85 to 6.95]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Fixed effects for treatment, prior antihyperglycemic medication, covariates for baseline A1C and baseline; Odds Ratio (OR) = 6.77, 95% CI 2-sided [3.46 to 13.24]

7. Secondary Outcome: Baseline 2-hour Post-prandial Glucose (2-hr PPG) Level
Description: Laboratory measurements were performed 120 minutes following the start of the administration of the meal for the Mixed Meal Tolerance Test (MMTT). Change from baseline in 2-hr PPG level at Week 26 data are presented in the following outcome measure.
Time Frame: Baseline
Population: Analysis population consisted of all randomized participants who had a baseline 2-hr PPG measurement.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 145 | 141 | 150
mg/dL | 260.32 (76.110) | 262.91 (78.189) | 256.21 (76.917)

8. Secondary Outcome: Change From Baseline in 2-hr PPG at Week 26
Description: The change from baseline is the Week 26 2-hr PPG minus the Week 0 2-hr PPG. Laboratory measurements were performed 120 minutes following the start of the administration of the meal for the MMTT. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study treatment and had a baseline 2-hr PPG measurement or at least 1 post-randomization 2-hr PPG measurement subsequent to at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 153 | 148 | 151
mg/dL | -64.15 [-74.34 to -53.96] | -62.45 [-72.91 to -51.98] | 4.88 [-6.15 to 15.92]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -69.03, 95% CI 2-sided [-83.24 to -54.83]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -67.33, 95% CI 2-sided [-81.73 to -52.93]

9. Secondary Outcome: Baseline Sitting Systolic Blood Pressure (SBP)
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. Change from baseline in SBP at Week 26 data are presented in the following outcome measure.
Time Frame: Baseline
Population: Analysis population consisted of all randomized participants who had a baseline SBP measurement.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 155 | 152 | 150
mmHg | 130.49 (13.511) | 129.67 (14.208) | 129.80 (14.464)

10. Secondary Outcome: Change From Baseline in SBP at Week 26
Description: The change from baseline is the Week 26 SBP minus the Week 0 SBP. Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study treatment and had a baseline SBP measurement or at least 1 post-randomization SBP measurement subsequent to at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 152 | 152
mmHg | -5.54 [-7.32 to -3.76] | -3.93 [-5.74 to -2.12] | -2.22 [-4.30 to -0.14]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.015, Constrained longitudinal data analysis — Nominal p-value; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -3.31, 95% CI 2-sided [-5.98 to -0.65]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.213, Constrained longitudinal data analysis; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -1.71, 95% CI 2-sided [-4.40 to 0.98]

11. Secondary Outcome: Baseline Sitting Diastolic Blood Pressure (DBP)
Description: Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. Change from baseline in DBP at Week 26 data are presented in the following outcome measure.
Time Frame: Baseline
Population: Analysis population consisted of all randomized participants who had a baseline DBP measurement.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 155 | 152 | 150
mmHg | 78.46 (8.117) | 78.53 (7.714) | 78.13 (7.458)

12. Secondary Outcome: Change From Baseline in DBP at Week 26
Description: The change from baseline is the Week 26 DBP minus the Week 0 DBP. Sitting blood pressure was measured in triplicate and the average of the measurements taken at a single assessment time was analyzed. Data presented exclude data following the initiation of rescue therapy.
Time Frame: Baseline and Week 26
Population: Analysis population consisted of all randomized participants who received at least 1 dose of study treatment and had a baseline DBP measurement or at least 1 post-randomization DBP measurement subsequent to at least 1 dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 156 | 152 | 152
mmHg | -2.52 [-3.65 to -1.40] | -1.10 [-2.24 to 0.05] | -0.72 [-2.05 to 0.60]
Statistical Analysis 1: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.039, Constrained longitudinal data analysis — Nominal p-value; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = -1.80, 95% CI 2-sided [-3.51 to -0.09]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority or Other; p = 0.669, Constrained longitudinal data analysis — Nominal p-value; [statistical method as in outcome 1, analysis 1]; Difference in least squares means = -0.37, 95% CI 2-sided [-2.09 to 1.35]

ADVERSE EVENTS:
Time Frame: Up to 54 weeks (+/- 3 days)
Description: Data presented below include data following the initiation of rescue therapy for the entire study (ie, all data after randomization, with no upper limit on the follow-up window for participants who discontinued study drug).
Arm/Group | Ertugliflozin 5 mg/Ertugliflozin 5 mg | Ertugliflozin 15 mg/Ertugliflozin 15 mg | Placebo/Metformin
Serious Adverse Events (participants affected / at risk) | 11/156 | 6/152 | 8/153
Other Adverse Events (participants affected / at risk) | 50/156 | 48/152 | 68/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg/Ertugliflozin 5 mg (N=156) | Ertugliflozin 15 mg/Ertugliflozin 15 mg (N=152) | Placebo/Metformin (N=153)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg/Ertugliflozin 5 mg (N=156) | Ertugliflozin 15 mg/Ertugliflozin 15 mg (N=152) | Placebo/Metformin (N=153)
Constipation (Gastrointestinal disorders) | 11 (11) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 5 (5) | 23 (26)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (4) | 12 (14)
Bronchitis (Infections and infestations) | 5 (5) | 1 (1) | 8 (9)
Nasopharyngitis (Infections and infestations) | 8 (8) | 11 (12) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 10 (11) | 9 (15)
Urinary tract infection (Infections and infestations) | 13 (15) | 10 (14) | 19 (30)
Vulvovaginal mycotic infection (Infections and infestations) | 12 (17) | 8 (11) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (4) | 6 (14) | 10 (23)
Headache (Nervous system disorders) | 6 (10) | 7 (9) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to Sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.